CLINICAL TRIAL: NCT01474317
Title: Performance of the G3 Blood Glucose Monitoring System With TATSU Strip
Brief Title: Study of an Investigational Glucose Meter System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ascensia Diabetes Care (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CTD-PRO-2010-009-01
Record Dates: First submitted 2011-11-16; First posted 2011-11-18 (Estimated); Results first posted 2013-01-03 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-01

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intended Users of the Monitoring System (Experimental): Untrained subjects with diabetes use the G3 investigational blood glucose monitoring system.
  Interventions: Device: G3 Investigational Blood Glucose Monitoring System

INTERVENTIONS:
Device: G3 Investigational Blood Glucose Monitoring System — Untrained subjects with diabetes perform self Blood Glucose (BG) tests with capillary fingerstick blood and AST of the palm using the G3 meter and an investigational sensor. Study staff test subject venous blood and all BG results are compared to a reference laboratory glucose method. Untrained subjects utilize some additional features of the meter using the User Guide and provide feedback.

SUMMARY:
The purpose of this study is to demonstrate that untrained subjects who have diabetes can operate the Investigational Blood Glucose Monitoring System (BGMS) and obtain valid glucose results.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 18 years of age and older
* Type 1 or type 2 diabetes
* Able to speak, read, and understand English
* Willing to complete all study procedures

Exclusion Criteria:

* Pregnancy
* Hemophilia or any other bleeding disorder
* Previously participated in a study using the G3 system
* Working for a medical laboratory, hospital or other clinical setting that involves training on and clinical use of blood glucose monitors.
* A condition, which in the opinion of the investigator, would put the person or study conduct at risk (reason for exclusion will be clearly documented by investigator or designee).
* Working for a competitive medical device company, or having an immediate family member or someone who is not a family member but is living within the household of someone who works for such a company.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2011-11; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bernstein, MD, FACE, Principal Investigator — Southwest Clinical Research Center; Michael Caswell, PhD, Principal Investigator — Consumer Product Testing Co.
Locations (2):
- United States (2):
  - Consumer Product Testing Co., Fairfield, New Jersey
  - Southwest Clinical Research Center, Santa Fe, New Mexico

RESULTS

PARTICIPANT FLOW:
Groups:
- Intended Users of the Monitoring System: Untrained subjects with diabetes use the G3 investigational blood glucose monitoring system.
  G3 Investigational Blood Glucose Monitoring System : Untrained subjects with diabetes perform self Blood Glucose (BG) tests with capillary fingerstick blood and AST of the palm using the G3 meter and an investigational sensor. Study staff test subject venous blood and all BG results are compared to a reference laboratory glucose method. Untrained subjects utilize some additional features of the meter using the User Guide and provide feedback.
Period: Overall Study
Arm/Group | Intended Users of the Monitoring System
Started | 226
Completed | 224
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Subject ineligible for study | 1

BASELINE CHARACTERISTICS:
Groups:
- Intended Users of the Monitoring System: Untrained subjects with diabetes use the G3 investigational blood glucose monitoring system. Of 226 subjects enrolled, 224 completed the study
  G3 Investigational Blood Glucose Monitoring System : Untrained subjects with diabetes perform self Blood Glucose (BG) tests with capillary fingerstick blood and AST of the palm using the G3 meter and an investigational sensor. Study staff test subject venous blood and all BG results are compared to a reference laboratory glucose method. Untrained subjects utilize some additional features of the meter using the User Guide and provide feedback.
Arm/Group | Intended Users of the Monitoring System
Number analyzed (Participants) | 224
Age, Continuous [Mean (Full Range); unit: years] — 224 subjects completed the study
  years | 54.4 [23 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 131
  Male | 93
Region of Enrollment [Number; unit: participants]
  United States | 224

OUTCOME MEASURES:

1. Primary Outcome: Percent of Self-Test Fingerstick Blood Glucose Results Within +/- 5to15mg/dL (<100mg/dL) or Within +/- 5to15% (>=100mg/dL) of Laboratory Glucose Method
Description: Untrained subjects with diabetes self-test fingerstick blood using an investigational Blood Glucose Monitoring System (BGMS). BGMS results are compared with capillary plasma BG results obtained with a Yellow Springs Instrument (YSI) Analyzer. YSI Analyzer BG results are used to calculate the number of BGMS results within +/- 5to15mg/dL (<100mg/dL YSI capillary plasma) or +/- 5to15% (>=100mg/dL YSI capillary plasma). Site staff tested in parallel after subjects.
Time Frame: 1 hour
Population: Blood data for three subjects were not evaluable because time defined in protocol was exceeded between meter test and blood sample preparation for reference method. 221 (224-3) blood test results were analyzed.
Measure: Number; unit: percentage of meter test results
Groups:
- Intended Users of the G3 Investigational BG Monitoring System: Untrained subjects with diabetes use the G3 investigational blood glucose monitoring system. Of 226 subjects enrolled, 224 completed the study.
  G3 Investigational Blood Glucose Monitoring System : Untrained subjects with diabetes perform self Blood Glucose (BG) tests with capillary fingerstick blood and AST of the palm using the G3 meter and an investigational sensor. Study staff test subject venous blood and all BG results are compared to a reference laboratory glucose method. Untrained subjects utilize some additional features of the meter using the User Guide and provide feedback.
Arm/Group | Intended Users of the G3 Investigational BG Monitoring System
Number analyzed (Participants) | 221
percentage of meter test results
  % within 15 mg/dL(<100 mg/dL BG) | 100
  % within 15% (>=100 mg/dL BG) | 98.9
  % within 12.5 mg/dL (<100 mg/dL BG) | 100
  % within 12.5% (>=100 mg/dL BG) | 98.4
  % within 10 mg/dL (<100 mg/dL BG) | 100
  % within 10% (>=100 mg/dL BG) | 95.6
  % within 5 mg/dL (<100 mg/dL BG) | 76.9
  % within 5% (>=100 mg/dL BG) | 78.6

2. Secondary Outcome: Percent of Glucose Results From Alternative Site Testing (AST) of the Palm Within +/- 15mg/dL (<75mg/dL) or Within +/- 20% (>=75mg/dL) of Laboratory Glucose Method
Description: Untrained subjects with diabetes self-test Alternative Site (AST) Palm blood using an investigational Blood Glucose Monitoring System (BGMS). BGMS AST results are compared with capillary plasma BG results obtained with a Yellow Springs Instrument (YSI) Analyzer. YSI capillary plasma BG results are used to calculate the number of AST BGMS results within +/- 15mg/dL (<75mg/dL YSI capillary plasma) or +/- 20% (>=75mg/dL YSI capillary plasma).
Time Frame: 1 hour
Population: Blood data for 3 subjects were not evaluable because time defined in protocol was exceeded between meter test and blood sample preparation for reference method. 221 (224-3) blood test results were analyzed.
Measure: Number; unit: percentage of meter test results
Arm/Group | Intended Users of the G3 Investigational BG Monitoring System
Number analyzed (Participants) | 221
percentage of meter test results
  % within 15 mg/dL (<75 mg/dL BG) | 100
  % within 20% (>=75 mg/dL BG) | 99.1

3. Secondary Outcome: Percent of Venous Blood Glucose Results Within +/- 5to15mg/dL (<75mg/dL) or Within +/- 5to20% (>=75mg/dL) of Laboratory Glucose Method
Description: Study staff tested subject venous blood using an investigational Blood Glucose Monitoring System (BGMS). Venous BGMS results are compared with venous plasma BG results obtained with a Yellow Springs Instrument (YSI) Analyzer. YSI venous plasma results are used to calculate the number of BGMS results within +/- 5to15mg/dL (<75mg/dL YSI venous plasma) or +/- 5to20% (>=75mg/dL YSI venous plasma).
Time Frame: 1 hour
Population: Venipuncture was unsuccessful for one subject. 223 (224-1) venous blood test results were analyzed.
Measure: Number; unit: percentage of meter test results
Arm/Group | Intended Users of the G3 Investigational BG Monitoring System
Number analyzed (Participants) | 223
percentage of meter test results
  % within 20% (>=75 mg/dL BG) | 100
  % within 15% (>=75 mg/dL BG) | 99.5
  %within 15 mg/dL (<75 mg/dL BG) | 100
  % within 12.5% (>=75 mg/dL BG) | 99.1
  % within 12.5 mg/dL (<75 mg/dL BG) | 100
  % within 10% (>=75 mg/dL BG) | 98.6
  % within 10 mg/dL (<75 mg/dL BG) | 100
  % within 5% (>=75 mg/dL BG) | 71.4
  % within 5 mg/dL (<75 mg/dL BG) | 83.3

4. Secondary Outcome: Number of Subjects Able to Perform Given Tasks Using Product Labeling for Instruction
Description: After reading the instructions for use, and without assistance from the study staff, subjects use the BGMS to utilize some of the additional features of the system. Study staff documents Yes or No 'Did the subject complete the task successfully?'
Time Frame: 1 hour
Measure: Number; unit: participants
Arm/Group | Intended Users of the G3 Investigational BG Monitoring System
Number analyzed (Participants) | 224
participants
  Mark a test result as 'Before Meal' | 208
  Set a reminder | 203
  Access BG trends | 215

ADVERSE EVENTS:
Arm/Group | Intended Users of the G3 Investigational BG Monitoring System
Serious Adverse Events (participants affected / at risk) | 0/224
Other Adverse Events (participants affected / at risk) | 4/224
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intended Users of the G3 Investigational BG Monitoring System (N=224)
Hypoglycemia (Endocrine disorders) | 3 (3) — Hypoglycemia events were non-serious (mild), non-device related, and anticipated.
Hyperglycemia (Endocrine disorders) | 1 (1) — Hyperglycemic event was non-serious (mild), non-device related, and anticipated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days